CLINICAL TRIAL: NCT05263583
Title: A Phase 2, Multicenter, Open Label Dose-ranging Study of Sepantronium Bromide in Patients With Relapsed/Refractory c-Myc Rearranged High-grade B-cell Lymphoma (HGBCL)
Brief Title: Sepantronium Bromide for the Treatment of High-grade B-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cothera Bioscience, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PC002-01
Record Dates: First submitted 2022-02-16; First posted 2022-03-02 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: High-grade B-cell Lymphoma; Burkitt Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphatic Diseases; Lymphoma, High-Grade; C-MYC/BCL2 Double-Hit High-Grade B-Cell Lymphoma; C-MYC/BCL6 Double-Hit High-Grade B-Cell Lymphoma; C-Myc Gene Rearrangement
Keywords: Relapsed/refractory
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphatic Diseases; Lymphoma, Non-Hodgkin; Recurrence | interventions — sepantronium

STUDY DESIGN:
Intervention Model Description: Dose range findings study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Cohort 1 will receive a dose of 3.6 mg/m2/day of sepantronium bromide
  Interventions: Drug: Sepantronium Bromide
- Cohort 2 (Experimental): Cohort 1 will receive a dose of 4.8 mg/m2/day of sepantronium bromide
  Interventions: Drug: Sepantronium Bromide
- Recommended Phase 2 Dose - Cohort 3 (Experimental): The recommended Phase 2 dose will be established based on the safety, pharmacokinetic and pharmacodynamic data from Cohort 1 and Cohort 2
  Interventions: Drug: Sepantronium Bromide

INTERVENTIONS:
Drug: Sepantronium Bromide — continuous intravenous infusion
  Other Names: PC-002

SUMMARY:
This is a multi-center Phase 2 study to determine the safety and efficacy of sepantronium bromide (SepB) in adult patients with relapsed or refractory high-grade B-cell lymphoma

DETAILED DESCRIPTION:
This is a multi-center, open label, dose-ranging Phase 2 study evaluating the safety and efficacy of SepB in patients with relapsed/refractory c-Myc rearranged HGBCL.

Cohorts of three patients will be enrolled at each dose level for SepB with expansion to six patients, if necessary, to assess toxicity.

Following the completion of 2 cycles of treatment of each cohort, an independent Data Monitoring Committee (DMC) will review the safety data to assess study drug related toxicities from the current cohort. Following this review, a decision will be made to continue dose escalation to the next dose level, to declare that a given dose level is the level of dose-limiting toxicity (DLT) or to further explore toxicity at the dose level in question by enrolling additional subjects to a maximum of six subjects at that level.

An additional 6 patients will be enrolled at the recommended Phase 2 dose (RP2D). The RP2D will be established on the basis of the maximally tolerated dose between the two specified dose levels as well as other relevant data, including clinical signals of activity, pharmacokinetic (PK) and pharmacodynamic (PD) data.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histologic diagnosis of c-Myc rearranged high-grade B-cell lymphoma
* Relapse or refractory disease after at least one previous line of therapy
* Measurable disease as defined by 2014 Lugano classification
* ECOG performance status of 0-2
* Acceptable coagulation parameters

Exclusion Criteria:

* Allogeneic transplant within 3 months
* Autologous transplant without resolution of post-transplant cytopenias
* Known CNS involvement
* Average QT/QTc interval duration > 450 msec
* Inadequate marrow, hepatic or renal function
* Unresolved Grade 2 or greater toxicities from prior anticancer therapy
* Radiotherapy within prior 4 weeks
* Requires systemic immunosuppressive therapy
* Positive for Hepatis B or Hepatis C
* Seropositive for HIV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability and recommended Phase 2 dose of sepantronium bromide | From time of signing informed consent through 30 days after the last dose of study drug, an average of 6 months
  Frequency, severity and relatedness of adverse events and the frequency of adverse events requiring discontinuation of study drug or dose reductions

SECONDARY OUTCOMES:
Overall response rate | From first dose through the last dose of study drug, an average of 6 months
  The ORR is defined as the percentage of participants who achieve either a Partial Response or Complete Response at any time during the treatment phase
Complete response rate | From first dose of study drug through the last dose of study drug, an average of 6 months
  Percentage of patients who experience a confirmed Complete Response at any time during the treatment phase
Duration of response | From first dose of study drug through to time of progression, an average of 6 months
  Time from the first documentation of a Complete Response or a Partial Response until the time to objective tumor progression
Clinical benefit rate | From first dose of study drug through the last dose of study drug, an average of 6 months
  Proportion of patients who achieve a Complete Response, Partial Response or Stable Disease during the treatment phase
Overall survival | From first dose of study drug through date of death, irrespective of cause, an average of 6 months
  The time from the first dose of study drug until death from any cause or date of last follow-up for living and lost to follow-up patients
Progression Free Survival | From first dose of study drug through relapse, disease progression or death due to any cause, an average of 12 months
  The time from first dose until relapse, disease progression or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Vernon Jiang, PhD, Study Director — Cothera Bioscience
Locations (11):
- China (6):
  - Beijing Cancer Hospital, Beijing
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Henan Cancer Hospital, Henan
  - Shanghai East Hospital, Pudong
  - Tianjin Cancer Hospital, Tianjin
  - Tongji Hospital, Wuhan
- South Korea (5):
  - Dong-A University Hospital, Busan
  - Inje University Haeundae Paik hospital, Busan
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St.Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.